CLINICAL TRIAL: NCT04033822
Title: Fast Track Pathway to Accelerated Cholecystectomy Versus Standard of Care for Acute Cholecystitis
Brief Title: Fast Track Pathway to Accelerated Cholecystectomy
Acronym: FAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: P.J. Devereaux (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Sponsor-Investigator, P.J. Devereaux, PHRI Perioperative and Digital Health Research Director, Population Health Research Institute
Organization: Population Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAST Pilot
Record Dates: First submitted 2019-02-04; First posted 2019-07-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cholecystitis; Cholecystectomy
Keywords: cholecystitis; cholecystectomy; accelerated surgery; feasibility study
MeSH Terms: conditions — Cholecystitis | interventions — Cholecystectomy

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trial, efficacy trial
Who Masked: Outcomes Assessor
Masking Description: allocation group will not be displayed. All personal identifying information will be removed and a computer generated participant ID will be used instead.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients randomized to the standard of care arm of the trial will not receive accelerated cholecystectomy surgery to correct cholecystitis. No services will be taken away but patients will continue with care as originally provided by the healthcare system.
- FAST Intervention (Experimental): Patients diagnosed with cholecystitis and randomized to the FAST intervention arm of the study will undergo surgery as soon as possible with a goal of surgery within 6 hours of diagnosis.
  Interventions: Procedure: cholecystectomy

INTERVENTIONS:
Procedure: cholecystectomy — If patients are randomized to the intervention arm of the study; said patient will undergo corrective cholecystectomy surgery to correct cholecystitis as soon as possible with a goal of surgery within 6 hours of diagnosis.
  Arms: FAST Intervention

SUMMARY:
More than 10% of Canadians have gallstones, and approximately 10% of these individuals will develop gallbladder inflammation related to gallstones, which is referred to as acute cholecystitis (AC). Patients with AC who do not have their gallbladder surgically removed have a 30% risk of serious complications that can lead to death. Surgery is the only definitive treatment for AC, however, there is controversy regarding the ideal timing of surgery. The two main approaches are early surgery (typically within 7 days of diagnosis) or delayed surgery (7 days to 6 weeks after diagnosis). Although preliminary evidence suggests that early surgery is associated with shorter hospital length of stay, lower risk for complications, and lower costs, practice varies widely regarding the timing of surgery. The limitations of the existing studies include small sample sizes, varied definitions of early versus delayed surgery, and an imbalance of risk between study groups. The proposed pilot study aims to inform the design of a large clinical trial that will compare the outcomes of patients with AC who receive accelerated surgery (i.e., as soon as possible with a goal of surgery within 6 hours of diagnosis) with those who receive standard care.

DETAILED DESCRIPTION:
The prevalence of gallstones is 10% and approximately 10% of patients develop acute cholecystitis (AC). AC prevalence increases with age and complications are as high as 30% in patients who do not undergo surgery, the only definitive treatment. There is controversy regarding ideal surgical timing. Previously, delayed surgery was thought to decrease bile duct injuries resulting from active inflammation. However, the state of persistent inflammation, hypercoagulability, and stress can cause medical complications such as myocardial injury. Chronic inflammation can lead to fibrosis, adhesions and higher chance of bile duct injuries during delayed surgery. There is also concern for recurrent AC episodes, recurrent pain, biliary pancreatitis, cholangitis or sepsis.

Recent studies suggest that early surgery may be associated with better outcomes, but practice remains variable, ranging anywhere from early surgery (<7 days) to delayed surgery (>7 days). Among >24,000 Ontarians with AC admitted to 106 hospitals, timing of cholecystectomy varied widely across sites. Only 58% of patients underwent surgery within 7 days. High volume hospitals were more likely to perform early surgery.17

Among 14,200 Ontarians with AC, a propensity score analysis demonstrated that early surgery was associated with less bile duct injury (relative risk (RR)=0.53, 95% confidence interval (CI) 0.31-0.90) and shorter length of hospital stay (LOS) (mean 1.9 days, 95% CI 1.7-2.1). Early surgery was less costly and more effective than delayed cholecystectomy.

Trials of surgical timing in patients with AC are limited. The largest randomized controlled trial (RCT) compared early and delayed surgery for AC only included 618 patients.9 Cholecystectomy was performed a median of 1 day after randomization in the early group compared to a median of 25 days in the delayed group. Duration of surgery and conversion rate to open surgery were similar in both groups. Early surgery was associated with less morbidity (11.8% vs. 34.4%, p<0.001), shorter LOS (5.4 vs. 10.0 days, p<0.001), and lower cost (€2919 vs. €4262, p<0.001).

Multiple meta-analyses have suggested that early surgery for AC is associated with fewer wound infections (RR 0.57; 95% CI 0.35-0.93) and have suggested a trend to fewer complications (RR 0.66; 95% CI 0.42-1.03). Limitations of these meta-analyses include studies with small sample sizes, few events, wide confidence intervals, and variation in the definition of early surgery. Finally, there is a lack of strong evidence to make definitive conclusions regarding impact of early surgery in AC, which has led to substantial variation in clinical practice.

AC initiates inflammatory, hypercoagulable, and stress states that can cause medical complications. Early surgical treatment will reduce the time patients are exposed to these harmful states and therefore may reduce the risk of complications. Furthermore, rapid surgery results in a shorter period of AC, which may impact hospital costs. The goal is to undertake a large multicentre RCT of the impact of accelerated surgery (goal within 6 hours of diagnosis) vs. usual timing of surgery in patients with AC on a composite outcome of major clinical and surgical complications at 90 days. "Standard of care", as described, is highly variable and depends on the surgeon and hospital practice patterns.

The main objective of this pilot study is to assess the feasibility of a large trial. The team hypothesizes that accelerated surgery for AC will improve clinical and surgical outcomes. A large RCT on this topic is needed for the following reasons: 1) time to surgery is a modifiable factor; 2) available data are encouraging, but not definitive; 3) there is variation in clinical practice across Ontario and internationally 4) the definition of early surgery has varied substantially across studies; 5) available data may be substantially underestimating the effect of timing of surgery because no trial has evaluated surgery within 6 hours of diagnosis; 6) high-quality evidence will modify clinical practice; and 7) implementation of accelerated surgery could save millions of healthcare dollars annually.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥45 years; or age ≥18 years and <45 years with at least one of the following co-morbidities: diabetes or chronic respiratory, cardiovascular, or renal disease;
2. Diagnosis of acute cholecystitis defined by the presence of at least 2 of the following:

   1. Abdominal pain in upper right quadrant,
   2. Murphy's sign,
   3. Leukocytosis >10 × 103/μl, or
   4. Oral temperature <36.5°C or >38°C;
3. Cholelithiasis (stones/sludge);
4. Ultrasound signs of cholecystitis;
5. Acute cholecystitis that requires surgery and is diagnosed during working hours;
6. Expected to require at least an overnight hospital admission after surgery; and
7. Provide written informed consent to participate in FAST.

Exclusion Criteria

1. Patients requiring emergent surgery or emergent interventions for another reason;
2. Patients whose therapeutic anticoagulation is not reversible;
3. Patients with a history of heparin-induced thrombocytopenia and current use of warfarin with an INR ≥1.5;
4. Pregnant patients;
5. Previous participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility (pertaining to patient recruitment) | 1 year
  Proportion of patients who are randomized into the trial.
Feasibility (pertaining to adherence to follow-up assessment) | 90 days post-randomization
  Proportion of patients with missed assessments and incomplete data variables
Feasibility (pertaining to patients who are randomized to Accelerated Care) | Within 6 hours after diagnosis of acute cholecystitis
  Proportion of patients who have surgery initiated within 6 hours of the diagnosis of acute cholecystitis among those randomly assigned to accelerated care.

SECONDARY OUTCOMES:
Hospital Length of Stay | 2 weeks
  Cumulative length of hospital stay related to acute cholecystitis
Proportion of patients who experience e a composite of Clinical Outcomes | 90 days after randomization
  Proportion of patients who experience: all-cause mortality, non-fatal sepsis, surgical site infection, pneumonia, Clostridium difficile-associated diarrhea, intra-abdominal abscess, bile duct injury, cystic duct stump leak, conversion to open surgery, intra-abdominal re-operation, intra-abdominal percutaneous or endoscopic re-intervention including placement of drain, embolization or Endoscopic Retrograde Cholangio-Pancreatography (ERCP), cholangitis, pancreatitis, myocardial injury, stroke, venous thromboembolism (VTE), new atrial fibrillation, congestive heart failure, new acute renal injury requiring dialysis and major bleeding.
Length of surgical procedure | 1 week
  Length of surgical procedure related to acute cholecystitis
Proportion of patients who experience acute kidney injury | 90 days after randomization
  Proportion of acute kidney injury events related to acute cholecystitis
Proportion of patients who are admitted to ICU within 90 days of randomization | 90 days after randomization
  Proportion of patients who are admitted to ICU related to acute cholecystitis
Number of hospital readmissions within 90 days of randomization | 90 days after randomization
  Number of hospital readmissions related to acute cholecystitis
Proportion of patients who experience peripheral arterial thrombosis within 90 days of randomization | 90 days after randomization
  Proportion of patients who experience peripheral arterial thrombosis related to acute cholecystitis
Proportion of patients who experience intra-operative cholangiogram | 1 day
  Rate of Cholangiogram related to acute cholecystitis
Subtotal cholecystectomy rate | 1 year
  Rate of cholecystectomies
Proportion of postoperative ileus | 2 weeks
  Proportion of postoperative ileus related to acute cholecystitis

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Kessler Borges PhD, M.D, Principal Investigator — Population Health Research Institute; Rahima Nenshi Msc, M.D, Principal Investigator — St. Joseph's Health Care London; PJ Devereaux PhD, M.D, Principal Investigator — Hamilton Health Sciences Corporation
Locations (4):
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Lawson Health Research Institute, London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borges FK, Nenshi R, Serrano PE, Engels P, Vogt K, Park LJ, Di Sante E, Vincent J, Tsiplova K, Devereaux PJ. Fast Track Pathway to Accelerated Cholecystectomy Versus Standard of Care for Acute Cholecystitis (FAST) pilot trial. Can J Surg. 2025 Apr 11;68(2):E122-E131. doi: 10.1503/cjs.016423. Print 2025 Mar-Apr. PMID 40216437